CLINICAL TRIAL: NCT01489111
Title: Efficacy and Safety of NNC 0129-0000-1003 During Surgical Procedures in Patients With Haemophilia A
Brief Title: Evaluating the Haemostatic Effect of NNC 0129-0000-1003 During Surgical Procedures in Subjects With Haemophilia A.
Acronym: pathfinder™3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NN7088-3860; U1111-1119-7326 (Other: WHO); 2011-001144-30 (EudraCT Number); 132215 (Other: JapicCTI)
Record Dates: First submitted 2011-11-23; First posted 2011-12-09 (Estimated); Results first posted 2020-01-21 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-07

CONDITIONS: Congenital Bleeding Disorder; Haemophilia A
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Surgery (Experimental)
  Interventions: Drug: turoctocog alfa pegol

INTERVENTIONS:
Drug: turoctocog alfa pegol — Bleeding preventive treatment administered i.v. before, during and after surgery. Individually adjusted doses.
  Other Names: NNC 0129-0000-1003

SUMMARY:
This trial is conducted globally. The aim of this trial is to evaluate the haemostatic effect of NNC 0129-0000-1003 during surgical procedures in subjects with haemophilia A.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities. (Trial-related activities are any procedure that would not have been performed during normal management of the subject.)
* Ongoing participation in the pathfinder™2 (NN7088-3859) or the pathfinderTM 4 (NN7088-3861) trial and having received greater than or equal to 5 doses of N8-GP
* Undergoing major surgery requiring daily monitoring of FVIII:C (FVIII activity) and wound status for at least 3 days
* The patient and/or Legally Acceptable Representative (LAR) is capable of assessing a bleeding episode, keeping an eDiary, capable of home treatment of bleeding episodes and otherwise capable of following the trial procedures

Exclusion Criteria:

* Known or suspected hypersensitivity to trial product including allergy to hamster protein or related products
* Previous withdrawal from the pathfinder™2 (NN7088-3859) or the pathfinderTM 4 (NN7088-3861) trial after administration of trial product, except interruption due to inclusion in this pathfinderTM 3 trial (NN7088-3860)
* The receipt of any investigational medicinal product (except N8-GP) within 30 days prior to enrolment into the trial. (For Brazil, only: Participation in a previous clinical trial within one year prior to screening for this trial (Visit 1), unless there is a direct benefit to the research subject, at the Investigator's discretion)
* FVIII inhibitors at least 0.6 BU (Bethesda Units)/mL at screening
* Previous arterial thrombotic events (e.g. myocardial infarction and intracranial thrombosis) or previous deep venous thrombosis or pulmonary embolism (as defined by available medical records)
* Immune modulating or chemotherapeutic medication
* Any disease (liver, kidney, inflammatory and mental disorders included) or condition which, according to the Investigator's judgement, could imply a potential hazard to the patient, interfere with trial participation or trial outcome
* Unwillingness, language or other barriers precluding adequate understanding and/or cooperation

Min Age: 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-08-03 (Actual); Primary Completion 2018-12-10 (Actual); Study Completion 2018-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (69):
- United States (19):
  - Novo Nordisk Investigational Site, Phoenix, Arizona
  - Novo Nordisk Investigational Site, Long Beach, California
  - Novo Nordisk Investigational Site, Sacramento, California
  - Novo Nordisk Investigational Site, Torrance, California
  - Novo Nordisk Investigational Site, Orlando, Florida
  - Novo Nordisk Investigational Site, Tampa, Florida
  - Novo Nordisk Investigational Site, Boise, Idaho
  - Novo Nordisk Investigational Site, Iowa City, Iowa
  - Novo Nordisk Investigational Site, New Orleans, Louisiana
  - Novo Nordisk Investigational Site, Baltimore, Maryland
  - Novo Nordisk Investigational Site, Newark, New Jersey
  - Novo Nordisk Investigational Site, Cincinnati, Ohio
  - Novo Nordisk Investigational Site, Portland, Oregon
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Charleston, South Carolina
  - Novo Nordisk Investigational Site, Nashville, Tennessee
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, Norfolk, Virginia
  - Novo Nordisk Investigational Site, Spokane, Washington
- Australia (3):
  - Novo Nordisk Investigational Site, Camperdown, New South Wales
  - Novo Nordisk Investigational Site, South Brisbane, Queensland
  - Novo Nordisk Investigational Site, Parkville, Victoria
- Novo Nordisk Investigational Site, Campinas, São Paulo, Brazil
- Novo Nordisk Investigational Site, Sofia, Bulgaria
- Croatia (2):
  - Novo Nordisk Investigational Site, Split
  - Novo Nordisk Investigational Site, Zagreb
- Denmark (2):
  - Novo Nordisk Investigational Site, Århus N
  - Novo Nordisk Investigational Site, København Ø
- France (4):
  - Novo Nordisk Investigational Site, Bron
  - Novo Nordisk Investigational Site, Le Kremlin-Bicêtre
  - Novo Nordisk Investigational Site, Nantes
  - Novo Nordisk Investigational Site, Paris
- Germany (6):
  - Novo Nordisk Investigational Site, Berlin
  - Novo Nordisk Investigational Site, Bonn
  - Novo Nordisk Investigational Site, Frankfurt/M.
  - Novo Nordisk Investigational Site, Hanover
  - Novo Nordisk Investigational Site, Homburg
  - Novo Nordisk Investigational Site, München
- Hungary (2):
  - Novo Nordisk Investigational Site, Budapest
  - Novo Nordisk Investigational Site, Debrecen
- Novo Nordisk Investigational Site, Tel Litwinsky, Israel
- Italy (3):
  - Novo Nordisk Investigational Site, Milan
  - Novo Nordisk Investigational Site, Udine
  - Novo Nordisk Investigational Site, Vicenza
- Japan (4):
  - Novo Nordisk Investigational Site, Kashihara-shi, Nara
  - Novo Nordisk Investigational Site, Shinjuku-ku, Tokyo
  - Novo Nordisk Investigational Site, Suginami-ku, Tokyo
  - Novo Nordisk Investigational Site, Tokyo
- Malaysia (2):
  - Novo Nordisk Investigational Site, Kuala Lumpur
  - Novo Nordisk Investigational Site, Selangor Darul Ehsan
- Netherlands (2):
  - Novo Nordisk Investigational Site, Groningen
  - Novo Nordisk Investigational Site, Rotterdam
- Novo Nordisk Investigational Site, Oslo, Norway
- Spain (2):
  - Novo Nordisk Investigational Site, Madrid
  - Novo Nordisk Investigational Site, Málaga
- Novo Nordisk Investigational Site, Malmo, Sweden
- Switzerland (3):
  - Novo Nordisk Investigational Site, Geneva
  - Novo Nordisk Investigational Site, Lausanne
  - Novo Nordisk Investigational Site, Zurich
- Taiwan (2):
  - Novo Nordisk Investigational Site, Changhua
  - Novo Nordisk Investigational Site, Taipei
- Turkey (Türkiye) (3):
  - Novo Nordisk Investigational Site, Adana
  - Novo Nordisk Investigational Site, Bornova-IZMIR
  - Novo Nordisk Investigational Site, Samsun
- United Kingdom (5):
  - Novo Nordisk Investigational Site, Basingstoke
  - Novo Nordisk Investigational Site, Cardiff
  - Novo Nordisk Investigational Site, London
  - Novo Nordisk Investigational Site, Oxford
  - Novo Nordisk Investigational Site, Sheffield

REFERENCES:
- [Result] Tosetto A, Neff A, Lentz SR, Santagostino E, Nemes L, Sathar J, Meijer K, Chowdary P, Shen C, Landorph A, Hampton K. Turoctocog alfa pegol provides effective management for major and minor surgical procedures in patients across all age groups with severe haemophilia A: Full data set from the pathfinder 3 and 5 phase III trials. Haemophilia. 2020 May;26(3):450-458. doi: 10.1111/hae.13980. Epub 2020 Apr 15. PMID 32293786
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 26 sites in 13 countries, as follows: Australia (1 site), Denmark (1 site), France (3 sites), Hungary (1 site), Israel (1 site), Italy (2 sites), Japan (2 sites), Malaysia (1 site), Netherlands (1 site), Switzerland (2 sites), Turkey (3 sites), United Kingdom (4 sites) and United States (4 sites).
Pre-assignment Details: 36 participants were screened and exposed to the trial product. A total of 53 surgeries were planned in these 36 participants and 49 surgeries were completed. The results are analysed and presented based on the number of surgeries instead of number of participants. Participants in this trial were also enrolled in the NN7088-3859 trial.
Units Other Than Participants: Surgeries
Groups:
- NNC 0129-0000-1003 (Turoctocog Alfa Pegol): Subjects (from trial NN7088-3859) undergoing major surgery received bleeding preventive treatment with turoctocog alfa pegol (N8-GP) before, during and after surgery. The trial product was administered as a slow bolus intravenous injection. Dosing was done at the investigators' discretion (except a fixed dose of 50 IU/kg at screening visit). The dose level of N8-GP during this trial was chosen following the coagulation factor 8 (FVIII) activity levels recommended by World Federation of Hemophilia (WFH) guidelines. The WFH guidelines for desired FVIII levels in major surgery are as follows: pre-surgery (day 0): 80-100%; post-surgery days 1-3: 60-80%; days 4-6: 40-60%; days 7-14: 30-50%. All subjects were treated with doses between 20-75 IU/kg for treatment of a bleeding episode. The maximum dose to be administered to a subject within 24 hours was 200 IU/kg. The total duration of the trial was 2-5 weeks. Upon completion of this trial, subjects returned to trial NN7088-3859.
Period: Overall Study
Arm/Group | NNC 0129-0000-1003 (Turoctocog Alfa Pegol)
Started | 36; 53 Surgeries
Completed | 35; 49 Surgeries
Not Completed | 1; 4 Surgeries
Not completed — Withdrawal criterion | 1

BASELINE CHARACTERISTICS:
Units Other Than Participants: Surgeries
Arm/Group | NNC 0129-0000-1003 (Turoctocog Alfa Pegol)
Number analyzed (Participants) | 36
Number analyzed (Surgeries) | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.6 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The number of partiipants enrolled were 36 while the number of planned surgeries were 53.
  Participants
    Female | 0
    Male | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The number of partiipants enrolled were 36 while the number of planned surgeries were 53.
  Participants
    Hispanic or Latino | 0
    Not Hispanic or Latino | 36
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The number of partiipants enrolled were 36 while the number of planned surgeries were 53.
  Participants
    American Indian or Alaska Native | 0
    Asian | 5
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 1
    White | 30
    More than one race | 0
    Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Haemostatic Effect During Surgery Evaluated by the Four-point Scale, Assessed by the Investigator/Surgeon at the Day of Surgery - Four-point Response Scale: Excellent, Good, Moderate or None
Description: Haemostatic effect during surgery was evaluated on a four-point response scale as 'none', 'moderate', 'good' and 'excellent'. This was assessed after completion of surgery (defined as "last stitch").
  Excellent: Better than expected/predicted in this type of procedure. Good: As expected in this type of procedure. Moderate: Less than optimal for the type of procedure but haemostatic response maintained without change of treatment regimen.
  None: Bleeding due to inadequate therapeutic response with adequate dosing, change of regimen required.
Time Frame: Assessed by the Investigator/surgeon at the day of surgery
Population: Full analysis set included all subjects exposed to the trial drug (N8-GP). 'Number Analyzed' = number of surgeries evaluated. 49 surgeries were evaluated in 35 participants.
Measure: Number; unit: Surgeries
Units Other Than Participants: Surgeries
Arm/Group | NNC 0129-0000-1003 (Turoctocog Alfa Pegol)
Number analyzed (Participants) | 35
Number analyzed (Surgeries) | 49
Surgeries
  Excellent | 25
  Good | 22
  Moderate | 2
  None | 0

2. Secondary Outcome: Average Consumption of N8-GP During Surgery
Description: Average consumption of N8-GP, during surgery is presented. The time during surgery is defined from 'knife to skin' until 'last stitch'.
Time Frame: During surgery, defined as the time from "knife to skin" until "last stitch"
Population: Full analysis set included all subjects exposed to the trial drug (N8-GP). 'Number Analyzed' = number of surgeries evaluated. N8-GP was administered during 1 surgery for 1 participant.
Measure: Number; unit: IU/kg
Units Other Than Participants: Surgeries
Arm/Group | NNC 0129-0000-1003 (Turoctocog Alfa Pegol)
Number analyzed (Participants) | 1
Number analyzed (Surgeries) | 1
IU/kg | 20.7 (0.0)

3. Secondary Outcome: Haemostatic Effect of N8-GP During the Post-operative Period Days 1-6
Description: Haemostatic effect during post-operative period days 1-6 as evaluated on a four-point response scale as 'none', 'moderate', 'good' and 'excellent'.
  Excellent: Better than expected/predicted in this type of procedure. Good: As expected in this type of procedure. Moderate: Less than optimal for the type of procedure but haemostatic response maintained without change of treatment regimen.
  None: Bleeding due to inadequate therapeutic response with adequate dosing, change of regimen required.
Time Frame: During the post-operative period, days 1-6
Population: Full analysis set included all subjects exposed to the trial drug (N8-GP). 'Number Analyzed' = number of surgeries evaluated. 2 surgeries with 2 bleeding episodes were evaluated in 35 participants.
Measure: Number; unit: bleeding episodes
Units Other Than Participants: bleeding episodes
Arm/Group | NNC 0129-0000-1003 (Turoctocog Alfa Pegol)
Number analyzed (Participants) | 35
Number analyzed (bleeding episodes) | 2
bleeding episodes
  Excellent | 0
  Good | 1
  Moderate | 0
  None | 0
  Missing | 1

4. Secondary Outcome: Haemostatic Effect of N8-GP During the Post-operative Period Days 7-14
Description: Haemostatic effect during post-operative period days 1-6 and days 7-14 was evaluated on a four-point response scale as 'none', 'moderate', 'good' and 'excellent'.
  Excellent: Better than expected/predicted in this type of procedure. Good: As expected in this type of procedure. Moderate: Less than optimal for the type of procedure but haemostatic response maintained without change of treatment regimen.
  None: Bleeding due to inadequate therapeutic response with adequate dosing, change of regimen required.
Time Frame: During the post-operative period, days 7-14
Population: as for outcome 3
Measure: Number; unit: bleeding episodes
Units Other Than Participants: bleeding episodes
Arm/Group | NNC 0129-0000-1003 (Turoctocog Alfa Pegol)
Number analyzed (Participants) | 35
Number analyzed (bleeding episodes) | 2
bleeding episodes
  Excellent | 1
  Good | 1
  Moderate | 0
  None | 0

5. Secondary Outcome: Average Consumption of N8-GP During the Post-operative Period Days 1-6
Description: Average consumption of N8-GP during post operative period days 1-6 is presented. Analysis population: Full analysis set included all subjects exposed to the trial drug (N8-GP) and completed surgery.
Time Frame: During the post-operative period, days 1-6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: IU/kg
Units Other Than Participants: Surgeries
Arm/Group | NNC 0129-0000-1003 (Turoctocog Alfa Pegol)
Number analyzed (Participants) | 35
Number analyzed (Surgeries) | 49
IU/kg | 33.0 (10.2)

6. Secondary Outcome: Incidence Rate of Inhibitors Against Factor VIII (FVIII) (≥0.6 BU/mL)
Description: Incidence rate of inhibitors is the number of newly developed inhibitors per surgery. Development of FVIII inhibitors was measured by a validated Nijmegen modified Bethesda assay. A positive inhibitor test was defined as ≥0.6 bethesda unit. Number of participants with inhibitors at the end of trial is presented.
Time Frame: during the trial (2-5 weeks)
Population: Safety analysis set (SAS) included all patients exposed to trial drug (N8-GP).
Measure: Number; unit: Participants
Arm/Group | NNC 0129-0000-1003 (Turoctocog Alfa Pegol)
Number analyzed (Participants) | 36
Participants | 0

7. Secondary Outcome: Estimated Blood Loss During Surgery
Description: The mean estimated blood loss following surgery is presented. Estimated blood loss (mL) was evaluated post surgery.
Time Frame: During surgery
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL
Units Other Than Participants: Surgeries
Arm/Group | NNC 0129-0000-1003 (Turoctocog Alfa Pegol)
Number analyzed (Participants) | 35
Number analyzed (Surgeries) | 49
mL | 322.6 (745.0)

8. Secondary Outcome: Number of Transfusions During the Post-operative Period Days 1-6
Description: Number of blood product transfusions (transfusion of red blood cells) during the post-surgery period, Days 1-6 is presented.
Time Frame: Post-operative period, days 1-6
Population: Full analysis set included all subjects exposed to the trial drug (N8-GP). 'Number Analyzed' = number of surgeries evaluated.
Measure: Number; unit: blood transfusions
Units Other Than Participants: Surgeries
Arm/Group | NNC 0129-0000-1003 (Turoctocog Alfa Pegol)
Number analyzed (Participants) | 35
Number analyzed (Surgeries) | 49
blood transfusions | 9

9. Secondary Outcome: Length of Stay in the Hospital
Description: Mean number of days stayed at the hospital during the trial.
Time Frame: During the trial (2-5 weeks)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: days
Units Other Than Participants: Surgeries
Arm/Group | NNC 0129-0000-1003 (Turoctocog Alfa Pegol)
Number analyzed (Participants) | 35
Number analyzed (Surgeries) | 49
days | 10.00 (8.9)

10. Secondary Outcome: Number of Days in Intensive Care
Description: Mean number of days in the intensive care due to surgery during the trial is presented.
Time Frame: During the trial (2-5 weeks)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: days
Units Other Than Participants: Surgeries
Arm/Group | NNC 0129-0000-1003 (Turoctocog Alfa Pegol)
Number analyzed (Participants) | 35
Number analyzed (Surgeries) | 49
days | 0.02 (0.14)

11. Secondary Outcome: Adverse Events Reported During the Trial Period
Description: Number of adverse event during the trial is presented. This includes events from the first trial related activity after the patient has signed the informed consent and until the end of trial (earliest at day 14).
Time Frame: During the trial (2-5 weeks)
Population: Safety analysis set (SAS) included all patients exposed to trial drug (N8-GP). 'Number Analyzed' = number of surgeries evaluated.
Measure: Number; unit: adverse events
Units Other Than Participants: Planned surgeries
Arm/Group | NNC 0129-0000-1003 (Turoctocog Alfa Pegol)
Number analyzed (Participants) | 36
Number analyzed (Planned surgeries) | 53
adverse events | 127

12. Secondary Outcome: Serious Adverse Events Reported During the Trial Period
Description: Number of serious adverse event during the trial is presented. This includes events from the first trial related activity after the patient has signed the informed consent and until the end of trial (earliest at day 14).
Time Frame: During the trial (2-5 weeks)
Population: as for outcome 11
Measure: Number; unit: serious adverse event
Units Other Than Participants: planned surgeries
Arm/Group | NNC 0129-0000-1003 (Turoctocog Alfa Pegol)
Number analyzed (Participants) | 36
Number analyzed (planned surgeries) | 53
serious adverse event | 5

ADVERSE EVENTS:
Time Frame: From the first trial related activity (day 0) after the patient has signed the informed consent until the end of trial (earliest at day 14).
Description: Adverse events were reported for the safety analysis set (SAS) which includes all subjects exposed to trial drug (N8-GP).
  As one of the objectives of the trial was to evaluate safety of N8-GP when used for prevention and treatment of bleeding throughout the surgical period, the adverse events are analysed based on the number (units) of surgeries rather than number of participants. Therefore 'the number at risk' in this adverse events section refers to the number of planned surgeries.
Arm/Group | NNC 0129-0000-1003 (Turoctocog Alfa Pegol)
All-Cause Mortality (participants affected / at risk) | 0/53
Serious Adverse Events (participants affected / at risk) | 4/53
Other Adverse Events (participants affected / at risk) | 30/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NNC 0129-0000-1003 (Turoctocog Alfa Pegol) (N=53)
Haemorrhage (Vascular disorders) | 1 (1)
Ischaemia (Vascular disorders) | 1 (1)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NNC 0129-0000-1003 (Turoctocog Alfa Pegol) (N=53)
Alanine aminotransferase increased (Investigations) | 3 (3)
C-reactive protein increased (Investigations) | 5 (5)
Constipation (Gastrointestinal disorders) | 11 (11)
Diarrhoea (Gastrointestinal disorders) | 3 (3)
Haemoglobin decreased (Investigations) | 5 (5)
Nausea (Gastrointestinal disorders) | 6 (6)
Post procedural inflammation (Injury, poisoning and procedural complications) | 3 (3)
Procedural pain (Injury, poisoning and procedural complications) | 5 (5)
Pyrexia (General disorders) | 4 (4)
Vomiting (Gastrointestinal disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-06): https://cdn.clinicaltrials.gov/large-docs/11/NCT01489111/Prot_SAP_000.pdf